CLINICAL TRIAL: NCT04159259
Title: Effect of Pea Fiber Supplementation on the Gut Microbiota and Host Metabolome and Proteome
Brief Title: Effect of Pea Fiber Supplementation on the Gut Microbiota and Host Metabolome and Proteome (FIB)
Acronym: FIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201812063
Record Dates: First submitted 2019-03-21; First posted 2019-11-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet intervention (Experimental): All participants will stay weight stable while undergoing 3 phases of a dietary intervention
  Interventions: Other: Low fiber diet; Other: Pea Fiber Bar

INTERVENTIONS:
Other: Low fiber diet — Participants will be provided with a low fiber diet in the form of packed out meals and snacks for 24 days in total (days 5-14 and days 36-49)
Other: Pea Fiber Bar — Participants will be provided with a low fiber diet plus 1-3 daily pea fiber bars from days 15-35
Other: Low fiber diet — Participants will return to the low fiber diet for days 36-49- this phase is the same as phase 1.

SUMMARY:
All subjects will complete a 49-day, multi-phase feeding study to evaluate the effect of pea fiber supplementation on gut community structure and features of host biological state (plasma proteome/ metabolome). Subjects will be asked to continue to consume their habitual diet (free diet phase) for 4 days prior to being provided with a diet high in saturated fat (HiSF) and low in fruits and vegetables (LoFV) in the form of packed-out meals and snacks to consume for the following 45 days. Ten days after starting to consume the HiSF-LoFV diet, subjects will supplement their diet with pea fiber for a total of 21 days; the energy contribution from the HiSF-LoFV diet will be reduced accordingly to maintain energy needs during this time. After completing the pea fiber supplementation phase of the study subjects will revert back to consuming the HiSF-LoFV only diet for the final 14 days. Stool, urine and blood will be sampled periodically throughout.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25.0-35.0 kg/m²
* Presence of B. vulgatus and B. thetaiotaomicron each at greater than 0.01% relative abundance

Exclusion Criteria:

* Previous bariatric surgery
* Significant organ system dysfunction (e.g. diabetes, severe pulmonary, kidney, liver, or cardiovascular disease)
* Cancer or cancer that has been in remission for less than 5 years
* Major psychiatric illness
* Inflammatory gastrointestinal disease
* Pregnant or lactating women
* Use of medications that are known to affect the study outcome measures
* Use of medications or supplements known to affect composition of the gut microbiota within the last 30 days (e.g. antibiotics)
* Bowel movements less than 3 times per week
* Vegans, vegetarians, and those with allergies, aversions, or sensitivities to foods provided in the study
* Persons that are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who the research team deems not an appropriate candidate for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in plasma lipid profile as assessed by the complete metabolic panel and lipid panel. | At screening, day 14, day 35, and day 49
  Blood will be drawn for the complete metabolic panel and lipid panel
Changes to the gut microbiota as assessed by established culture independent methods, as well as LC-QTOF Mass-Spectometry (MS) and LC-QQQ MS and GC-MS | stool samples will be collected from the screening visit through the final day of the 49-day intervention
  Frequent stool samples will be collected throughout the entire study
Changes in urine proteomes and metabolomes as assessed by liquid chromatography | Daily or every other day first-morning urine samples will be collected from day 1 to day 49 of the study
  First morning urine samples will be collected periodically throughout the study
Changes in plasma proteomes and metabolomes as assessed by liquid chromatography | Fasted blood draws will be collected on days 1, 14, 21, 28, 35, and 49 of the study
  fasting blood draws will be collected periodically throughout the study
Change in hemoglobin A1c (HbA1c) in response to the dietary intervention | At screening, day 14, day 35, and day 49
  Blood will be drawn for the HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Tara Wilmot, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided